CLINICAL TRIAL: NCT05983367
Title: A Randomized Phase 2 Study of Ompenaclid Versus Placebo in Combination With FOLFIRI Plus Bevacizumab in Patients With Previously Treated RAS Mutant Advanced or Metastatic Colorectal Cancer
Brief Title: A Study to Investigate Ompenaclid Combined With FOLFIRI Plus Bevacizumab in Advanced/Metastatic Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inspirna, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGX-202-002
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Metastatic Colon Cancer
Keywords: Metastatic colon cancer; KRAS colon cancer; CRC advance cancer; malignant colorectal tumor; RAS mutant colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: randomized 1:1
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ompenaclid + FOLFIRI + Bevacizumab (Experimental): Ompenaclid (RGX-202-01) 3000mg PO (tablets) BID; Irinotecan: 180 mg/m2 over 90 minutes concurrently with folinic acid 400 mg/m2 over 2 hours, followed by 5-FU 2400 mg/m2 over 46 hours, on Days 1 and 15 of each 28-day cycle. Bevacizumab: 5 mg/kg on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Ompenaclid; Drug: Bevacizumab; Drug: FOLFIRI regimen
- Placebo + FOLFIRI + Bevacizumab (Placebo Comparator): Placebo (tablets) PO + Irinotecan: 180 mg/m2 over 90 minutes concurrently with folinic acid 400 mg/m2 over 2 hours, followed by 5-FU 2400 mg/m2 over 46 hours, on Days 1 and 15 of each 28-day cycle. Bevacizumab: 5 mg/kg on Days 1 and 15 of each 28-day cycle.
  Interventions: Drug: Placebo; Drug: Bevacizumab; Drug: FOLFIRI regimen

INTERVENTIONS:
Drug: Ompenaclid — Ompenaclid (RGX-202-01)
  Other Names: RGX-202-01
  Arms: Ompenaclid + FOLFIRI + Bevacizumab
Drug: Placebo — Placebo
  Arms: Placebo + FOLFIRI + Bevacizumab
Drug: Bevacizumab — Bevacizumab
Drug: FOLFIRI regimen — FOLFIRI regimen (irinotecan 180 mg/m2 over 90 minutes concurrently with folinic acid 400 mg/m2 over 2 hours, and then 5-FU 2400 mg/m2 over 46 hours on Days 1 and 15 of each 28-day cycle)

SUMMARY:
The purpose of this study is to measure tumor response to treatment with ompenaclid (RGX-202-01) in patients with previously treated RAS mutant advanced or metastatic CRC. All patients will receive treatment with FOLFIRI and bevacizumab. In addition, patients will be randomized to receive either ompenaclid 3000 mg BID or matching placebo (herein referred to as Study Drug). Each treatment cycle is 28 days in duration.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind placebo-controlled study of ompenaclid or matching placebo (Study Drug) in combination with standard-of-care FOLFIRI plus bevacizumab as background therapy in patients with previously treated RAS mutant advanced or metastatic CRC. Randomization will be stratified by whether or not the patient received prior treatment with bevacizumab or an EMA-approved biosimilar. Written informed consent must be obtained prior to initiating any screening activities, except where patients have agreed to the use of previously available tests completed within 28 days of the planned first dose of Study Drug, e.g., computed tomography (CT)/magnetic resonance imaging (MRI) scans. Screening for study eligibility must be completed within 28 days prior to first dose of Study Drug. Patients who are determined to be eligible, based on Screening assessments, will be randomized in the study, and receive their first dose of Study Drug on Cycle 1, Day 1. A treatment cycle is 28 days in duration. Patients will be randomized in a 1:1 ratio to receive oral administration of the five 600-mg tablets BID of ompenaclid or matching placebo (Study Drug). The intravenous FOLFIRI dose and schedule for all patients will be irinotecan 180 mg/m2 over 90 minutes concurrently with folinic acid 400 mg/m2 over 2 hours,followed by 5-FU 2400 mg/m2 over 46 hours, on Days 1 and 15 of each 28-day cycle. The bevacizumab dose of 5 mg/kg will be administered intravenously on Days 1 and 15 of each 28-day cycle. During treatment, patients will attend study center visits and have study evaluations performed as detailed in the Schedule of Events (Table 1-1). All routine study visits are to be conducted on an outpatient basis. Patients may continue to receive Study Drug until the development of PD, or another discontinuation criterion is met, including unacceptable toxicity, voluntary withdrawal from treatment, or closure of the study by the Sponsor; no maximum duration of therapy has been set. After discontinuation of the Study Drug, patients will complete an End of Treatment (EOT) visit within 21 days after their last dose of Study Drug. Safety follow-up is to be conducted by telephone 30 days (+/- 3 days) after their last dose of Study Drug and longer if drug-related AEs have not resolved at that time. Patients and/or their health care providers will also be contacted by telephone approximately every 90 days for information on evidence of PD in settings in which discontinuation of Study Drug was for reasons other than PD, such as an adverse event (AE) or investigator discretion, and/or for assessment of survival status (tumor measurements as specified in the protocol are not required after the EOT visit). This extended follow-up for disease status and survival after discontinuation of the Study Drug may continue until the target number of disease progression events have been observed or for 12 months after the patient's EOT visit, whichever is later. The End of Study for a given patient is defined as the date of the last extended follow-up disease/survival status, or until death, withdrawal of consent, loss to follow-up, or study closure, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria

1. Advanced disease, defined as cancer that is either metastatic or locally advanced and unresectable and for which additional radiation therapy or other locoregional therapies are not considered feasible.
2. Progression of disease after receiving only 1 prior regimen considered standard of care for CRC in the advanced/metastatic setting, and it must have been an oxaliplatin containing regimen. Patients who have mismatch repair deficiency/ high microsatellite instability (dMMR/MSI-H) CRC must have also received prior treatment with pembrolizumab or a Food and Drug Administration (FDA)/European Union (EU)-approved programmed cell death protein 1 (PD-1)/ programmed death-ligand 1 (PD-L1) inhibitor. Patients may have received prior treatment with bevacizumab or an European Medicines Agency (EMA) approved biosimilar. Patients who developed metastatic CRC within 12 months of completion of adjuvant oxaliplatin and 5-FU based therapy are also eligible.
3. Histologic or cytologic evidence of a malignant colorectal tumor of adenocarcinoma or poorly differentiated histology that is laboratory-confirmed to be RAS mutant. Confirmation of RAS mutant status by liquid biopsy is acceptable only if the tumor sample is not available and the liquid biopsy was performed before initiation of the patient's prior treatment regimen. Patients who convert to RAS mutant status after initially having documented wild-type histology are not eligible.
4. Disease that is measurable by standard imaging techniques by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. For patients with prior radiation therapy, measurable lesions must be outside of any prior radiation field(s), unless disease progression has been documented at that disease site subsequent to radiation.
5. At least 18 years old.
6. ECOG performance score ≤ 1.
7. Adequate baseline organ function, as demonstrated by the following:

   1. Calculated creatinine clearance > 60 mL/min per institutional standard.
   2. Serum albumin ≥ 2.5 g/dL.
   3. Bilirubin ≤ 1.5 x institutional upper limit of normal range (ULN).
   4. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x institutional ULN; patients with hepatic metastases may have AST and ALT ≤ 5 x institutional ULN.
   5. Absolute neutrophil count (ANC) ≥1.5x109/L.
   6. Hemoglobin ≥ 8 g/dL and no red blood cell (RBC) transfusions during the prior 14 days.
   7. Platelet count ≥ 100 x 109/L and no platelet transfusions during the prior 14 days.
8. If not taking warfarin (or similar vitamin K inhibitor) the following values are required: international normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 x ULN and either partial thromboplastin time or activated partial thromboplastin time (PTT or aPTT) ≤ 1.5 x ULN. Patients on warfarin (or similar vitamin K inhibitor) may be included if on a stable dose with a therapeutic INR < 3.5.
9. Left ventricular ejection fraction (LVEF) x 45% as determined by either echocardiography (ECHO) or multigated acquisition (MUGA) scanning.
10. Woman of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 2 weeks prior to treatment.
11. Men and WOCBP must agree to use acceptable contraceptive methods for the duration of time on the study and continue to use acceptable contraceptive methods for at least 6 months from the last dose of bevacizumab or 2 months after the last dose of ompenaclid, whichever is longer.
12. Provides signed informed consent prior to initiation of any study-specific procedures or treatment.
13. Able to adhere to the study visit schedule and other protocol requirements, including follow-up for survival assessment

Exclusion Criteria:

1. Persistent clinically significant toxicities (Grade ≥ 2) from previous anticancer therapy. Excluded are Grade 2 chemotherapy-related neuropathy and alopecia which are permitted and Grade 2 laboratory abnormalities if they are not associated with symptoms, are not considered clinically significant by the Investigator, or can be managed with available medical therapies.
2. CRC with histology (or component of histology) consistent with small cell, neuroendocrine, or squamous carcinoma, or lymphoma.
3. Received treatment with chemotherapy, external-beam radiation, or other systemic anticancer therapy within 14 days prior to study therapy administration (42 days for prior nitrosourea or mitomycin-C).
4. Received treatment with an investigational systemic anticancer agent within 5 half lives of the investigational systemic therapy or within 28 days, whichever is shorter prior to Study Drug administration.
5. Has an additional active malignancy that may confound the assessment of the study endpoints. Patients with a past cancer history with substantial potential for recurrence must be discussed with the Medical Monitor before study entry. Patients with the following concomitant neoplastic diagnoses are eligible: non-melanoma skin cancer, carcinoma in situ (including transitional cell carcinoma, cervical intraepithelial neoplasia, and melanoma in situ), organ-confined prostate cancer with no evidence of progressive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | From randomization until development of radiographic disease progression (estimated up to 24 months).
  ORR is defined as the proportion of patients achieving a best overall response (BOR) of complete response (CR) or partial response (PR) per the investigators using RECIST version 1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization until development of radiographic disease progression or death due to any cause, whichever comes first (estimated up to 24 months).
  PFS is defined as the time from the date of randomization to the date of objectively determined progressive disease (PD) per the investigators using RECIST version 1.1 or death from any cause, whichever occurs first.
Overall Survival (OS) | From randomization until death due to any cause (estimated up to 36 months).
  OS is defined as the time from the date of randomization to the date of death from any cause.
Duration of Response (DoR) | From randomization until development of radiographic disease progression or death due to any cause, whichever comes first (estimated up to 24 months).
  DoR is defined as the time from the date of objectively determined PR or CR (whichever status is recorded first) to the date of PD per the investigators using RECIST version 1.1 or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | From randomization until development of radiographic disease progression (estimated up to 24 months).
  DCR is defined as the proportion of patients achieving a BOR of CR, PR, or stable disease (SD).
Frequency of Adverse Events (AEs) | From the signing of informed consent until 30 days (+/- 3 days) after the last dose of study drug. (estimated up to 24 months).
  Percentage of patients with treatment-emergent AEs (TEAE).
Pharmacokinetics of ompenaclid | At Cycle 1 day 15 and Cycle 2 day 15 (each cycle is 28 days in length).
  Steady state concentration
Exploratory biomarkers that may correlate with efficacy outcomes | At baseline
  CKB levels identified in baseline tumor samples

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Takahashi, MD, Study Director — Inspirna, Inc.
Locations (28):
- Belgium (8):
  - Imelda Ziekenhuis, Bonheiden, Antwerpen
  - Universite Catholique de Louvain (UCL) - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital
  - Institut Jules Bordet, Anderlecht
  - Antwerp University Hospital, Antwerp
  - UZ Brussel, Brussels
  - Grand Hoptial De Charleroi, Charleroi
  - UZ Leuven, Leuven
  - CHU de Liège University hospital in Liège, Liège
- France (8):
  - CHU Nantes -hopital hotel Dieu, Nantes, Loire-Atlantique
  - CHU Hôpital Jean Minjoz, Besançon
  - Centre Georges-François Leclerc, Dijon
  - Institut Paoli-Calmettes, Marseille
  - Groupe Hospitalier Paris Saint Joseph - Oncologie, Paris
  - Hopital Prive des Cotes d'Armor, Plérin
  - Institut de Cancerologie de l'Ouest, Saint-Herblain
  - Institut Gustave Roussy, Villejuif
- Spain (12):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Puerta de Hierro Majadahonda, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Clinico De Valencia, Valencia
  - Hospital Clinico Universitario De Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided